CLINICAL TRIAL: NCT04950829
Title: Evaluation of Leveling and Alignment Time and the Periodontal Status in Patients With Severe Upper Crowding Treated by Flapless Corticotomy-assisted Self-ligating Brackets in Comparison With Conventional or Self-Ligating Brackets Alone
Brief Title: Efficacy and Periodontal Parameters in Self-ligating Brackets Alone or With Corticotomy vs Conventional Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-05-2021
Record Dates: First submitted 2021-06-19; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Crowding of Anterior Maxillary Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional brackets (Active Comparator): Patients will receive an orthodontic treatment using conventional brackets until achieving appropriate alignment of the upper anterior teeth.
  Interventions: Device: Conventional brackets
- Self-ligating brackets (Experimental): Patients will receive an orthodontic treatment using self-ligating brackets until achieving appropriate alignment of the upper anterior teeth.
  Interventions: Device: Self-ligating brackets
- 3- Self-Ligating brackets with fapless corticotomy (Experimental): Patients will receive an orthodontic treatment using self-ligating brackets with corticotomy until achieving appropriate alignment of the upper anterior teeth.
  Interventions: Procedure: Self-Ligating Brackets with flapless corticotomy

INTERVENTIONS:
Device: Conventional brackets — These brackets are used in a conventional way, where the orthodontist used to apply elastic parts to engage the arch to the slot of the brackets.
  Arms: Conventional brackets
Device: Self-ligating brackets — These brackets do not need to use elastic parts to engage the arch to the brackets. The orthodontist can use sliding caps to open and close the slots of these brackets.
  Arms: Self-ligating brackets
Procedure: Self-Ligating Brackets with flapless corticotomy — These brackets do not need to use elastic parts to engage the arch to the brackets. The orthodontist can use sliding caps to open and close the slots of these brackets.
  Flapless corticotomy will be performed in order to stimulate acceleration in tooth movement during the orthodontic treatment in this group only.
  Arms: 3- Self-Ligating brackets with fapless corticotomy

SUMMARY:
Patients who have severe crowding on the upper jaw that requires two first premolars extraction will be enrolled in this trial. The different types of brackets, such as self-ligating brackets and conventional brackets, and the various acceleration methods, such as corticotomy, have different effects on the orthodontic treatment time and the periodontal tissues. So, this study will assess and compare the overall leveling and aligning time and the changes in periodontal indices between patients with severe crowding, treating with self-ligating brackets associated with flapless corticotomy versus conventional brackets alone versus self-ligating brackets alone.

There are three groups:

The first group (control group): the patients in this group will be treated using conventional brackets alone.

The second group (Experimental group): the patients in this group will be treated using self-ligating brackets alone.

The third group (Experimental group): the patients in this group will be treated using self-ligating brackets associated with flapless corticotomy.

DETAILED DESCRIPTION:
The prolonged duration of the treatment period can cause many problems such as caries and periodontal diseases. The oral environment is considered a suitable environment for many germs and microorganisms to grow. Any increase in the percentage of these germs predisposes to the occurrence of dental and periodontal problems.

Several studies have used various procedures and many types of brackets to accelerate dental movement in order to reduce treatment time.

Orthodontic treatment using different devices usually contributes to change the nature of the oral environment and its contents of microorganisms Many bracket systems have been used, such as the conventional brackets and self-ligating brackets. The use of self-ligating brackets has increased significantly in recent years. The absence of wired or elastic elements may cause less accumulation of plaque.

ELIGIBILITY:
Inclusion Criteria:

* Sever crowding greater than 6 mm on the upper jaw in which orthodontic treatment requires extraction of two upper premolars.
* The Little's Index of Irregularity is more than 7 mm.
* Good oral health (plaque Index is less or equal to 1).
* Class I or class II (ANB ≤ 5) or class III (ANB ≥ 0).
* Overbite is between 0-4 mm.
* No skeletal constriction on the upper jaw.
* No congenitally missing or extracted teeth (except for the third molars).

Exclusion Criteria:

* Any systemic diseases affect teeth movement.
* Any congenital syndromes or cleft lip and palate.
* Bad oral health.
* The patient is not committed to periodic follow-up times.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Duration of teeth alignment | This will be measured immediately at the end of the alignment stage; this is expected to be within 180 to 200 days
  The number of days required to finish the alignment stage of upper teeth will be calculated from the beginning of treatment till the end of the alignment stage (i.e. teeth alignment is achieved)

SECONDARY OUTCOMES:
The change in the plaque index. | T0: immediately before applying the fixed appliance; T1: after 1 month; T2: after 2 months, T3: after 3 months, T4: after 6 months
  Assessment will be achieved using a gingival probe according to Silness and Loe (1964).
  A. (0) = No plaque. B. (1) = A film of plaque stick to the free gingival margin and adjacent area of the tooth.
  C. (2) = Moderate accretion of soft deposits on the tooth and gingival margin or within the gingival pocket.
  D. (3) = Abundance of soft material on the tooth and gingival margin and/or within the gingival pocket.
The change in the gingival index | T0: immediately before applying the fixed appliance; T1: after 1 month; T2: after 2 months, T3: after 3 months, T4: after 6 months
  Assessment will be achieved using a gingival probe according to Silness and Loe (1964).
  A. (0) = Normal gingiva. B. (1) = Mild inflammation: minor change in color, slight oedema. No bleeding on probing.
  C. (2) = Moderate inflammation: redness, oedema and glazing and bleeding on probing.
  D. (3) = Sever inflammation: marked redness and oedema, ulceration, and tendency to spontaneous bleeding
The change in papillary bleeding index. | T0: immediately before applying the fixed appliance; T1: after 1 month; T2: after 2 months, T3: after 3 months, T4: after 6 months
  Assessment will be achieved using a gingival probe according to Muhlemann (1977).
  A. (0) = No bleeding. B. (1) = A single discreet bleeding point appears. C. (2) = Several isolated bleeding points or a single fine line of blood appears.
  D. (3) = The interdental triangle fills with blood shortly after probing. E. (4) = Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
The change in the probing depth | T0: immediately before applying the fixed appliance; T1: after 1 month; T2: after 2 months, T3: after 3 months, T4: after 6 months
  Assessment will be achieved using a gingival probe according to Miller (1985) It will be measured clinically as the distance from the free gingival margin to the gingival sulcus.

CONTACTS AND LOCATIONS:
Overall Officials: Heba M AL-Ibrahim, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental; Mohammad Y Hajeer, Study Chair — Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Issam Khoury, DDS,MSc,PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergamo AZ, Nelson-Filho P, Romano FL, da Silva RA, Saraiva MC, da Silva LA, Matsumoto MA. Gingival crevicular fluid volume and periodontal parameters alterations after use of conventional and self-ligating brackets. J Orthod. 2016 Dec;43(4):260-267. doi: 10.1080/14653125.2016.1221214. Epub 2016 Sep 8. PMID 27607519
- [Background] Chhibber A, Agarwal S, Yadav S, Kuo CL, Upadhyay M. Which orthodontic appliance is best for oral hygiene? A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2018 Feb;153(2):175-183. doi: 10.1016/j.ajodo.2017.10.009. PMID 29407494
- [Background] Pandis N, Vlachopoulos K, Polychronopoulou A, Madianos P, Eliades T. Periodontal condition of the mandibular anterior dentition in patients with conventional and self-ligating brackets. Orthod Craniofac Res. 2008 Nov;11(4):211-5. doi: 10.1111/j.1601-6343.2008.00432.x. PMID 18950317
- [Background] Cozzani M, Ragazzini G, Delucchi A, Mutinelli S, Barreca C, Rinchuse DJ, Servetto R, Piras V. Oral hygiene compliance in orthodontic patients: a randomized controlled study on the effects of a post-treatment communication. Prog Orthod. 2016 Dec;17(1):41. doi: 10.1186/s40510-016-0154-9. Epub 2016 Dec 19. PMID 27891568
- [Background] Mulla Issa FHK, Mulla Issa ZHK, Rabah AF, Hu L. Periodontal parameters in adult patients with clear aligners orthodontics treatment versus three other types of brackets: A cross-sectional study. J Orthod Sci. 2020 Feb 12;9:4. doi: 10.4103/jos.JOS_54_17. eCollection 2020. PMID 32166083
- [Background] Lombardo L, Ortan YO, Gorgun O, Panza C, Scuzzo G, Siciliani G. Changes in the oral environment after placement of lingual and labial orthodontic appliances. Prog Orthod. 2013 Sep 11;14:28. doi: 10.1186/2196-1042-14-28. PMID 24326120